CLINICAL TRIAL: NCT00098878
Title: SCOTROC 4: A Prospective, Multicentre, Randomised Trial Of Carboplatin Flat Dosing Vs Intrapatient Dose Escalation In First Line Chemotherapy Of Ovarian, Fallopian Tube And Primary Peritoneal Cancers
Brief Title: Carboplatin in Treating Patients With Stage IC-IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SCOTTISH-SCOTROC-4; CDR0000396778 (Registry Identifier: PDQ (Physician Data Query)); EU-20402; ISRCTN47645935 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register))
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-07

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin

INTERVENTIONS:
Drug: carboplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This randomized phase III trial is comparing different doses of carboplatin to see how well they work in treating patients with stage IC, stage II, stage III, or stage IV ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of patients with stage IC-IV ovarian epithelial, fallopian tube, or primary peritoneal cancer treated with flat-dose vs intra-patient dose-escalated carboplatin as first-line chemotherapy.

Secondary

* Compare the toxic effects of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare overall clinical response rate and CA 125 response in patients treated with these regimens.
* Compare overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive a flat dose of carboplatin on day 1.
* Arm II: Patients receive intra-patient dose-escalated carboplatin on day 1. In both arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each treatment course, and then at 2 months post-chemotherapy.

Patients are followed every 2 months for 2 years, every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 1,300 patients (650 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cancer*

  * Stage IC-IV disease
  * Peritoneal carcinomatosis* (ovarian-type) must not be a mucin-secreting tumor
  * Stage IC patients must have malignant cells in ascitic fluid or peritoneal washings, tumor on the surface of the ovary, or preoperative capsule rupture NOTE: * Histologic confirmation of a primary source in the ovary is not required.
* If biospy is not available, cytology showing an adenocarcinoma is allowed provided the following criteria is met:

  * Patient has a pelvis (ovarian) mass AND all of the following:

    * Omental cake or other metastasis is larger than 2 cm in the upper abdomen and/or regional lymph node metastasis irrespective of size OR stage IV disease
    * Serum CA 125/CEA ratio > 25 or barium enema (or colonoscopy) and gastroscopy (or radiological examination of the stomach) are negative for the presence of a primary tumor and normal mammography within 6 weeks prior to study randomization
* Initial cytoreductive laparotomy or biopsy required within the past 8 weeks

  * Cytoreductive surgery may or may not have been successful during staging laparotomy
* No mixed mesodermal tumors
* No borderline ovarian tumors or tumors termed "possibly malignant"
* No adenocarcinoma of unknown origin, if histologically confirmed to be a mucin-secreting tumor
* Considered unsuitable for or unwilling to receive platinum-taxane combination therapy
* No concurrent endometrial cancer

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN

Renal

* Creatinine clearance ≥ 30 mL/min

  * Obstructive hydronephrosis as a cause of borderline (i.e., creatinine clearance 30-45 mL/min) renal function must be treated before study entry

Cardiovascular

* No hypertension
* No ischemic heart disease
* No myocardial infarction within the past 6 months
* No congestive heart failure

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No symptomatic peripheral neuropathy ≥ grade 2
* No uncontrolled infection
* No other severe and/or uncontrolled medical condition
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy
* No other concurrent cytotoxic chemotherapy until progressive disease occurs

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2004-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Toxicity
Quality of life
Clinical overall response rate and CA125 response
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Stanley B. Kaye, MD, FRCP, Study Chair — Royal Marsden NHS Foundation Trust
Locations (88):
- Australia (21):
  - Sydney Heamatology and Oncology Clinics, Hornsby, New South Wales
  - Lismore Base Hospital, Lismore, New South Wales
  - Institute of Oncology at Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Tamworth Base Hospital, Tamworth, New South Wales
  - Manning Base Hospital, Taree, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Wentworthville, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Townsville Hospital, Douglas, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Ballarat Oncology and Haematology Services, Ballarat, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Royal Women's Hospital, Carlton, Victoria
  - Monash Medical Center - Clayton Campus, Clayton, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Mercy Hospital for Women, Heidelberg, Victoria
  - Murray Valley Private Hospital and Cancer Treatment Centre, Wodonga, Victoria
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Wellington Cancer Centre, Wellington
- United Kingdom (63):
  - Furness General Hospital, Barrow in Furness, England
  - Royal United Hospital, Bath, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Royal Blackburn Hospital, Blackburn, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Bradford Royal Infirmary, Bradford, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Broomfield Hospital, Broomfield, England
  - Queen's Hospital, Burton-on-Trent, England
  - Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Derbyshire Royal Infirmary, Derby, England
  - Dorset County Hospital, Dorchester, England
  - Russells Hall Hospital, Dudley, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Hereford Hospitals NHS Trust, Hereford, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Ipswich Hospital, Ipswich, England
  - Airedale General Hospital, Keighley, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Liverpool Women's Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - University College of London Hospitals, London, England
  - Guy's Hospital, London, England
  - St. Georges, University of London, London, England
  - Hammersmith Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Kings Mill Hospital, Nottinghamshire, England
  - George Eliot Hospital, Nuneaton, England
  - Whiston Hospital, Prescot Merseyside, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Royal Marsden - Surrey, Sutton, England
  - Taunton and Somerset Hospital, Taunton Somerset, England
  - South Warwickshire Hospital, Warwick, Warwickshire, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Weston General Hospital, Weston-super-Mare, England
  - Worcester Royal Hospital, Worcester, England
  - Worthing Hospital, Worthing, England
  - Yeovil District Hospital, Yeovil - Somerset, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Dumfries & Galloway Royal Infirmary, Dumfries, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Gartnavel General Hospital, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - West Wales General Hospital, Carmarthen, Wales
  - South West Wales Cancer Institute, Swansea, Wales